CLINICAL TRIAL: NCT06002607
Title: Pilot Randomized Controlled Trial of Shorter Versus Extended Course of Antibiotic Therapy for Necrotizing Soft Tissue Infections
Brief Title: Shorter Versus Extended Course of Antibiotic Therapy for Necrotizing Soft Tissue Infections
Status: Recruiting | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Areg Grigorian, Assistant Clinical Professor, Surgery, University of California, Irvine
Other Study IDs: 2826
Record Dates: First submitted 2023-07-11; First posted 2023-08-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Necrotizing Soft Tissue Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biochemical procalcitonin on admission and daily for up to 7 days or after source control has been achieved.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Short course of antibiotics: Patients assigned to a 48-hour course of antibiotics. As the current standard of care, the antibiotics used in this treatment are Clindamycin, Vancomycin, Piperacillin-Tazobactam; these antibiotics may be administered combined or individually, based on individualized patient treatment. The specific choice of antibiotic therapy will not be dictated by the study protocol but by the attending surgeon taking care of the patient
  Interventions: Other: Antibiotic duration (short course)
- Long course of antibiotics: Patients assigned to a 7 day course of antibiotics. As the current standard of care, the antibiotics used in this treatment are Clindamycin, Vancomycin, Piperacillin-Tazobactam; these antibiotics may be administered combined or individually, based on individualized patient treatment. The specific choice of antibiotic therapy will not be dictated by the study protocol but by the attending surgeon taking care of the patient
  Interventions: Other: Antibiotic duration (extended course)

INTERVENTIONS:
Other: Antibiotic duration (short course) — The patient will be enrolled in a 48-hour course of antibiotics.
  Groups: Short course of antibiotics
Other: Antibiotic duration (extended course) — The patient will be enrolled in a 7 day course of antibiotics.
  Groups: Long course of antibiotics

SUMMARY:
Necrotizing soft tissue infection (NSTI) is a devastating disease that results in a high rate of in-hospital complications and despite advances in critical care, wound care, and early intervention, NSTI continues to be associated with a mortality rate of nearly 30%. The antibiotics used in this treatment are Clindamycin, Vancomycin, Piperacillin Tazobactam; these antibiotics may be administered combined or individually, based on individualized patient treatment. Although one of the tenets of management for NSTI is early broad-spectrum intravenous antibiotics (listed above), the duration of antibiotics needed is not well defined. Currently, there exists wide variation in the duration of antibiotics for NSTI ranging between 2-16 days. The objective of this study is to evaluate the safety of a shorter course of antibiotics hypothesizing that a short duration of antibiotics for 48-hours after source-control is achieved will have similar risk of morbidity and mortality compared to a 7-day course of antibiotics post source control. A second aim of this study will be to identify if serum procalcitonin levels/ratio correspond to resolution of systemic infection in patients with NSTI.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety of a shorter course of antibiotics hypothesizing that a short duration of antibiotics for 48-hours after source-control is achieved will have similar risk of morbidity and mortality compared to a 7-day course of antibiotics post source control. The proposed shortened duration is considered within standard of care as the IDSA suggests 48-72 hours of antibiotics after source control, however this was due mostly to expert opinion until a recent single-center study using historical controls demonstrated a 48-hour duration of antibiotics to be safe. A second aim of this study will be to identify if serum procalcitonin levels/ratio correspond to resolution of systemic infection in patients with NSTI. This pilot study may help limit use of antibiotics which are associated with both cost and significant adverse events including antimicrobial resistance and clostridium difficile infections. In addition, the data would support grant submission of a larger, multi-center study with sufficient power to demonstrate the safety profile and potential benefits of a shorter duration of antibiotics, which has been shown to be beneficial in previous large surgical infection studies.

Specific Aims:

Aim#1: Establish the safety of an abbreviated course (48 hours after source control) compared to a prolonged (7 days after source control) course of antibiotics in terms of in-hospital mortality.

Aim#2: Compare the incidence of hospital length of stay and in-hospital complications including unplanned return to the operating room, ventilator days, and antibiotic associated complications (e.g., clostridium difficile infection) in the two comparison groups: abbreviated (48-hours) and prolonged antibiotics (7-days) after source control.

Aim#3: Identify a critical threshold of biochemical procalcitonin or a % decrease in procalcitonin from the initial procalcitonin obtained upon admission that suggests resolution of systemic infection in patients with NSTI. This will be done by obtaining a serum procalcitonin upon admission and daily for up to 7 days from admission or once source control has been achieved.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age or older with all following criteria:
* Presenting to the Emergency Department with history, exam and/or imaging concerning NSTI, AND
* Patients who undergo consultation by the Emergency General Surgery service, AND
* Patients included must have skin or soft tissue findings consistent with NSTI (erythema, crepitus, or pain out of proportion to exam), AND
* Systemic signs of infection including fever (temperature >38.0°C) or leukocytosis (≥11,000 peripheral white cells per cubic millimeter), AND
* Patients who undergo excisional debridement and/or amputation to achieve source control.

Exclusion Criteria:

* Pregnant patients
* Prisoners
* Patients with bacteremia upon admission
* Patients unable to provide consent (including no legally authorized representative)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of Necortizing Soft Tissue Infection who undergo consultation by the Emergency General Surgery service.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety of the antibiotic course duration | Through study completion, an average of 1 year
  In-hospital complications
Mortality rate | Through study completion, an average of 1 year
  In-hospital mortality

SECONDARY OUTCOMES:
Age | Baseline, pre-intervention/procedure/surgery
  Age in years
Sex | Baseline, pre-intervention/procedure/surgery
  Sex (male/female)
BMI (body mass index) | Baseline, pre-intervention/procedure/surgery
  Body mass index (weight and height will be combined to report BMI in kg/m^2)
Blood Pressure | Baseline, pre-intervention/procedure/surgery
  Blood Pressure (mmHg)
Heart Rate | Baseline, pre-intervention/procedure/surgery
  Heart rate (beats/minute)
Respiratory rate | Baseline, pre-intervention/procedure/surgery
  Respiratory rate (breaths/minute)
Temperature | Baseline, pre-intervention/procedure/surgery
  Temperature (Fahrenheit)
Comorbidities | Baseline, pre-intervention/procedure/surgery
  Comorbidities (e.g., diabetes, hypertension, cirrhosis, chronic kidney disease, etc.)
Transfusion requirements | Baseline, pre-intervention/procedure/surgery
  Number of Packed Red Blood Cells transfused measured in milliliters
NSTI location | Baseline, pre-intervention/procedure/surgery
  Anatomical location of soft tissue infection
Operations | Through study completion, an average of 1 year
  Number of surgical procedures
Serum concentration of procalcitonin | Upon admission and daily blood sample for 7 days
  Procalcitonin ng/mL
Serum concentration of white blood cell | Through study completion, an average of 1 year
  White blood cell count cells per microliter (cells/μL)
Serum concentration of hemoglobin | Through study completion, an average of 1 year
  Hemoglobin grams/deciliter
Serum concentration of sodium | Through study completion, an average of 1 year
  Sodium millimoles per liter (mmol/L)
Serum concentration of C-reactive protein | Through study completion, an average of 1 year
  C-reactive protein milligrams/liter
Serum concentration of glucose | Through study completion, an average of 1 year
  Glucose milligrams/deciliter
Serum concentration of creatinine | Through study completion, an average of 1 year
  Creatinine milligram/deciliter
Total hospital length of stay | Through study completion, an average of 1 year
  Total days of hospital stay
Total intensive care unit (ICU) | Through study completion, an average of 1 year
  Total days of ICU stay
Total ventilator days | Through study completion, an average of 1 year
  Total days of ventilation support for the patient

CONTACTS AND LOCATIONS:
Overall Officials: Areg Grigorian, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No
The overall study results will be listed on Clinicaltrials.gov

REFERENCES:
- [Background] Yilmazlar T, Ozturk E, Alsoy A, Ozguc H. Necrotizing soft tissue infections: APACHE II score, dissemination, and survival. World J Surg. 2007 Sep;31(9):1858-1862. doi: 10.1007/s00268-007-9132-1. PMID 17610007
- [Background] Childers BJ, Potyondy LD, Nachreiner R, Rogers FR, Childers ER, Oberg KC, Hendricks DL, Hardesty RA. Necrotizing fasciitis: a fourteen-year retrospective study of 163 consecutive patients. Am Surg. 2002 Feb;68(2):109-16. PMID 11842952
- [Background] Hefny AF, Eid HO, Al-Hussona M, Idris KM, Abu-Zidan FM. Necrotizing fasciitis: a challenging diagnosis. Eur J Emerg Med. 2007 Feb;14(1):50-2. doi: 10.1097/01.mej.0000228447.48276.7b. PMID 17198329
- [Background] Stevens DL, Bisno AL, Chambers HF, Dellinger EP, Goldstein EJ, Gorbach SL, Hirschmann JV, Kaplan SL, Montoya JG, Wade JC; Infectious Diseases Society of America. Practice guidelines for the diagnosis and management of skin and soft tissue infections: 2014 update by the Infectious Diseases Society of America. Clin Infect Dis. 2014 Jul 15;59(2):e10-52. doi: 10.1093/cid/ciu444. PMID 24973422
- [Background] Schuetz P, Albrich W, Mueller B. Procalcitonin for diagnosis of infection and guide to antibiotic decisions: past, present and future. BMC Med. 2011 Sep 22;9:107. doi: 10.1186/1741-7015-9-107. PMID 21936959
- [Background] Becker KL, Nylen ES, White JC, Muller B, Snider RH Jr. Clinical review 167: Procalcitonin and the calcitonin gene family of peptides in inflammation, infection, and sepsis: a journey from calcitonin back to its precursors. J Clin Endocrinol Metab. 2004 Apr;89(4):1512-25. doi: 10.1210/jc.2002-021444. No abstract available. PMID 15070906
- [Background] Faraklas I, Yang D, Eggerstedt M, Zhai Y, Liebel P, Graves G, Dissanaike S, Mosier M, Cochran A. A Multi-Center Review of Care Patterns and Outcomes in Necrotizing Soft Tissue Infections. Surg Infect (Larchmt). 2016 Dec;17(6):773-778. doi: 10.1089/sur.2015.238. Epub 2016 Nov 11. PMID 27834617
- [Background] Terzian WTH, Nunn AM, Call EB, Bliss SE, Swinarska JT, Rigdon J, Avery MD, Hoth JJ, Miller PR 3rd. Duration of Antibiotic Therapy in Necrotizing Soft Tissue Infections: Shorter is Safe. Surg Infect (Larchmt). 2022 Jun;23(5):430-435. doi: 10.1089/sur.2022.011. Epub 2022 Apr 22. PMID 35451883
- [Background] May AK, Talisa VB, Wilfret DA, Bulger E, Dankner W, Bernard A, Yende S. Estimating the Impact of Necrotizing Soft Tissue Infections in the United States: Incidence and Re-Admissions. Surg Infect (Larchmt). 2021 Jun;22(5):509-515. doi: 10.1089/sur.2020.099. Epub 2020 Aug 21. PMID 32833599